CLINICAL TRIAL: NCT02320461
Title: Estudo Longitudinal de Saúde do Adulto
Brief Title: Estudo Longitudinal de Saúde do Adulto (Brazilian Longitudinal Study of Adult Health )
Acronym: ELSA-Brasil
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, MSchmidt, Associate Professor, Federal University of Rio Grande do Sul
Other Study IDs: 01.06.0010.00
Record Dates: First submitted 2014-12-16; First posted 2014-12-19 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Diabetes Mellitus; Cardiovascular Diseases
Keywords: diabetes mellitus; cardiovascular diseases; cohort studies; hypertension; obesity; smoking; social class
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases; Hypertension; Obesity; Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Frozen serum and urine samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The Brazilian Longitudinal Study of Adult Health (ELSA-Brasil) aims to contribute with relevant information regarding the development and progression of clinical and subclinical chronic diseases, particularly cardiovascular diseases and diabetes. The investigators enrolled 15,105 civil servants from predefined universities or research institutes. Baseline assessment (2008-2010) included detailed interviews and measurements to assess social and biological determinants of health, as well as various clinical and subclinical conditions related to diabetes, cardiovascular diseases and mental health. For the ascertainment of incident events, annual telephone surveillance is being conducted since 2009, and a second visit of interviews and exams is under way (2012-2014). Long-term biological sample storage is provided for sera, plasma, urine and DNA. Baseline data is available for analyses, and collaboration via specific research proposals directed to study investigators is welcome.

This multicenter study is chaired by a steering committee, made up of the coordinators and vice-coordinators of each of the six centers. No individual center coordinates the study. The six institutions listed in the contact details all sponsor the study.

DETAILED DESCRIPTION:
Full details of the study have been published in the American Journal of Epidemiology (http://aje.oxfordjournals.org/content/early/2012/01/10/aje.kwr294.full) and the International Journal of Epidemiology (http://ije.oxfordjournals.org/content/early/2014/02/27/ije.dyu027.abstract), as listed in the References here. Both articles are available in full text for download without charge.

ELIGIBILITY:
Inclusion Criteria:

* age 35-74 years,
* active or retired employees of the institutions involved or affiliated institutions.

Exclusion Criteria:

* current or recent (<4 months prior to the first interview) pregnancy,
* intention to quit work at the institution in the near future,
* severe cognitive or communication impairment and,
* if retired, residence outside each center´s corresponding metropolitan area.

Ages: 35 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ELSA-Brasil is a cohort study of 15,105 civil servants. All active or retired employees of the six institutions (and, in a few instances, also of related educational or health institutions), of both sexes, and with ages between 35 and 74 years, were eligible for the study. The six institutions, located in three different Brazilian regions, are: the Federal Universities of Bahia, Espirito Santo, Minas Gerais and Rio Grande do Sul, the University of Sao Paulo and the Oswaldo Cruz Foundation.
Sampling Method: Non-Probability Sample
Enrollment: 15105 (Actual)
Dates: Start 2008-08; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Diabetes mellitus (Incident cases) | 6 years
  Incident cases
Myocardial infarction (Incident cases) | 6 years
  Incident cases

CONTACTS AND LOCATIONS:
Overall Officials: Estela M Aquino, MD, Principal Investigator — Federal University of Bahia; José G Mill, MD, Principal Investigator — Federal University of Espirito Santo; Sandhi M Barreto, MD, Principal Investigator — Universidade Federal da Minas Gerais; Rosane H Griep, DSc, Principal Investigator — Fundação Oswaldo Cruz; Paulo A Lotufo, MD, Principal Investigator — University of Sao Paulo; Maria I Schmidt, MD, Principal Investigator — Federal University of Rio Grande do Sul

REFERENCES:
- [Background] Aquino EM, Barreto SM, Bensenor IM, Carvalho MS, Chor D, Duncan BB, Lotufo PA, Mill JG, Molina Mdel C, Mota EL, Passos VM, Schmidt MI, Szklo M. Brazilian Longitudinal Study of Adult Health (ELSA-Brasil): objectives and design. Am J Epidemiol. 2012 Feb 15;175(4):315-24. doi: 10.1093/aje/kwr294. Epub 2012 Jan 10. PMID 22234482
- [Background] Schmidt MI, Duncan BB, Mill JG, Lotufo PA, Chor D, Barreto SM, Aquino EM, Passos VM, Matos SM, Molina Mdel C, Carvalho MS, Bensenor IM. Cohort Profile: Longitudinal Study of Adult Health (ELSA-Brasil). Int J Epidemiol. 2015 Feb;44(1):68-75. doi: 10.1093/ije/dyu027. Epub 2014 Feb 27. PMID 24585730
- [Derived] Birck MG, Almeida-Pititto B, Janovsky CCPS, Goulart AC, Santos IS, Teixeira PFDS, Sgarbi JA, Barreto SM, Duncan BB, Schmidt MI, Lotufo PA, Bensenor IM. Thyroid-Stimulating Hormone and Thyroid Hormones and Incidence of Diabetes: Prospective Results of the Brazilian Longitudinal Study of Adult Health (ELSA-BRASIL). Thyroid. 2022 Jun;32(6):694-704. doi: 10.1089/thy.2021.0533. Epub 2022 May 24. PMID 35473396
- [Derived] Riboldi BP, Luft VC, Bracco PA, de Oliveira Cardoso L, Molina MDC, Alvim S, Giatti L, Schmidt MI, Duncan BB. The inflammatory food index and its association with weight gain and incidence of diabetes: Longitudinal Study of Adult Health (ELSA-Brasil). Nutr Metab Cardiovasc Dis. 2022 Mar;32(3):675-683. doi: 10.1016/j.numecd.2021.12.022. Epub 2022 Jan 6. PMID 35123853
- [Derived] Drehmer M, Odegaard AO, Schmidt MI, Duncan BB, Cardoso LO, Matos SMA, Molina MDCB, Barreto SM, Pereira MA. Brazilian dietary patterns and the dietary approaches to stop hypertension (DASH) diet-relationship with metabolic syndrome and newly diagnosed diabetes in the ELSA-Brasil study. Diabetol Metab Syndr. 2017 Feb 13;9:13. doi: 10.1186/s13098-017-0211-7. eCollection 2017. PMID 28228848
- [Derived] Drehmer M, Pereira MA, Schmidt MI, Del Carmen B Molina M, Alvim S, Lotufo PA, Duncan BB. Associations of dairy intake with glycemia and insulinemia, independent of obesity, in Brazilian adults: the Brazilian Longitudinal Study of Adult Health (ELSA-Brasil). Am J Clin Nutr. 2015 Apr;101(4):775-82. doi: 10.3945/ajcn.114.102152. Epub 2015 Jan 21. PMID 25833975
- See also: Public website of the study — http://www.elsa.org.br/